CLINICAL TRIAL: NCT04980872
Title: A Multicenter, Open-label, Phase 2, Extension Trial to Study the Long-term Safety in Participants With PROS or Proteus Syndrome Who Are Currently Being Treated With Miransertib in Other Studies
Brief Title: A Study of the Safety and Tolerability in Participants With PIK3CA-related Overgrowth Spectrum or Proteus Syndrome Who Are Being Treated With Miransertib (MK-7075) in Other Studies (MK-7075-006)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7075-006; MK-7075-006 (Other: MSD); 2022-500689-87-00 (Registry Identifier: EU CT); 2021-001369-19 (EudraCT Number)
Record Dates: First submitted 2021-07-23; First posted 2021-07-28 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: PIK3CA-Related Overgrowth Spectrum (PROS)/Proteus Syndrome (PS)
Keywords: ARQ 092; ArQule; AKT; mTOR; PIK3CA; PROS; Proteus; Overgrowth; Congenital malformations; MOSAIC
MeSH Terms: conditions — Hereditary Sensory and Autonomic Neuropathies; Proteus Infections; Congenital Abnormalities | interventions — Miransertib

STUDY DESIGN:
Intervention Model Description: Multicenter
Masking Description: None (Open-label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Miransertib (Experimental): Participants with either PROS or PS receive miransertib orally once daily between 5 and 35 mg/m^2 based on prior approved dosing for up to 96 cycles. A cycle is 28 days long.
  Interventions: Drug: Miransertib

INTERVENTIONS:
Drug: Miransertib — Miransertib capsules administered orally either 1 hour before or 2 hours after a meal.
  Other Names: MK-7075; ARQ 092

SUMMARY:
This is a study of the safety and tolerability of oral miransertib (MK-7075) administered to participants at least 2 years of age with phosphatidylinositol-4,5-bisphosphate 3-kinase catalytic subunit alpha (PIK3CA)-related overgrowth spectrum (PROS) or Proteus Syndrome (PS). This is an extension of other miransertib studies (MK-7075-002 [NCT03094832] or ArQule CU/EAP [NCT03317366]), and may also enroll participants who are approved for MK-7075-002 but have not yet started miransertib therapy.

ELIGIBILITY:
Inclusion Criteria:

* Has PROS or PS and has been screened in Study MK-7075-002 (or has been approved by the Sponsor to screen for MK-7075-002) or is currently being treated with miransertib as part of Study MK-7075-002 (NCT03094832) or ArQule's CU/EAP (NCT03317366)
* For males, agrees to be abstinent from heterosexual intercourse or use contraception unless confirmed to be azoospermic during the study period and for ≥90 days after the last dose of study intervention
* For females, is not pregnant or breastfeeding, and is either not a participant of childbearing potential (POCBP) or is a POCBP and is abstinent or uses a highly effective method of contraception

Exclusion Criteria:

* Has previously discontinued miransertib due to related SAEs or other intolerance of miransertib
* Has received other investigational agents, if any, that were administered between leaving Study MK-7075-02 or ArQule's CU/EAP and entering this trial
* Is receiving systemic inhibitors of the mechanistic target of rapamycin (mTOR) pathway (eg, sirolimus, everolimus)
* Is receiving immunosuppressive therapies
* Is receiving continuous high dose steroids

Ages: 2 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-11-02 (Actual); Primary Completion 2030-02-07 (Estimated); Study Completion 2030-02-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants experiencing a Serious Adverse Event (SAE) | Up to approximately 94 months
  An SAE is defined as any untoward medical occurrence associated with the use of a drug in a participant, whether or not considered drug related. An SAE can therefore be any such event that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalizations, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is considered by the investigator to be an important medical event.
Number of participants discontinuing study treatment due to an Adverse Event (AE) | Up to approximately 90 months
  An AE is defined as any untoward medical occurrence associated with the use of a drug in a participant, whether or not considered drug related. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product and does not imply any judgment about causality.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (11):
- United States (5):
  - Children's Healthcare of Atlanta - Egleston Hospital ( Site 0107), Atlanta, Georgia
  - Boston Children's Hospital ( Site 0089), Boston, Massachusetts
  - Cincinnati Children's Hospital Medical Center-Hematology ( Site 0102), Cincinnati, Ohio
  - Texas Children's Hospital ( Site 0104), Houston, Texas
  - Seattle Children's Hospital ( Site 0103), Seattle, Washington
- Australia (2):
  - John Hunter Hospital ( Site 0203), Newcastle, New South Wales
  - Bundaberg Base Hospital ( Site 0202), Bundaberg, Queensland
- Hospital Araújo Jorge ( Site 0801), Goiânia, Goiás, Brazil
- Italy (2):
  - Fondazione Policlinico Universitario Agostino Gemelli ( Site 0052), Rome, Lazio
  - Ospedale Pediatrico Bambino Gesù-Centro Trials ( Site 0087), Rome, Roma
- Great Ormond Street Hospital ( Site 0701), London, London, City of, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Oncology Clinical Trials Information — http://merckoncologyclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26218&tenant=MT_MSD_9011